CLINICAL TRIAL: NCT03007186
Title: Glucose Monitoring During Threatening Preterm Birth With Particular Focus on Insulin Sensitivity and Glucose Tolerance in Patients With and Without Gestational Diabetes Mellitus
Brief Title: Glucose Monitoring During Threatening Preterm Birth in Patients With and Without Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Lara Linsenmeier, Principal Investigator, Medical University of Vienna
Other Study IDs: 1102/2016
Record Dates: First submitted 2016-12-19; First posted 2017-01-02 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Diabetes, Gestational; Insulin Sensitivity; PreTerm Birth; Glucose Intolerance During Pregnancy; Glucocorticoids
Keywords: Blood glucose monitoring; Glucose tolerance; HbA1C; Insulin; Betamethasone
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case group: The oral glucose tolerance test that these women undergo in pregnancy between 24+0 and 28+0 showed pathological measurements.
- Control group: The oral glucose tolerance test of these women showed no pathological measurements.

SUMMARY:
This study aims to show whether the hyperglycaemic phases following a treatment with glucocorticoids, as well as blood measurements correlated to high blood glucose levels and insulin resistance, vary significantly between patients with and without gestational diabetes mellitus.

DETAILED DESCRIPTION:
BACKGROUND:

The therapy with glucocorticoids for fetal lung maturation in the case of threatening preterm birth is an long existing part of the obstetric routine procedures. Under this therapy it should not be forgotten, that glucocorticoids can lead to a decrease of the maternal insulin sensitivity as well as they can cause an impaired maternal glucose tolerance.

Therefore a threatening preterm birth as well as the including medical therapy do challenge the glucose metabolism of mother and child.

Gestational diabetes mellitus (GDM) is one of the most common complications during pregnancy, and the numbers are on the rise. GDM is characterized through an insulin resistance during the pregnancy.

High blood glucose level during pregnancy or labour can cause complications like a fetal hypoglycaemia right after birth.

METHODS:

This study includes pregnant women with and without gestational diabetes who are medicated with betamethasone due to threatening preterm birth.

In this study the blood glucose measurements of one week, as well as the measurements of HbA1C, Insulin and Blood Glucose from a blood draw one week after the lung maturation therapy will be considered.

ELIGIBILITY:
Inclusion Criteria:

* female
* gestational age between 23+0 and 34+6
* an oral glucose tolerance test was made and attests a healthy glucose tolerance (control group) a gestational diabetes mellitus (case group)
* threatening preterm birth

Exclusion Criteria:

* missing consent to participate
* age under 18 years
* age over 50 years
* preexistent diabetes (type 1 or 2)
* apparent disease of the thyroid gland
* infectious diseases as HIV or Hepatitis C
* insulin dependent gestational diabetes mellitus

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All participating patients will be pregnant women with a threatening preterm birth admitted to the department of feto-maternal health and obstetrics of the AKH Vienna.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-10; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Blood glucose measurements | Seven days after betamethasone medication.
  The patient measures their blood glucose level six times a day for seven days. The times of the measurements are before and one hour after every meal.

SECONDARY OUTCOMES:
HbA1C | One week after the medication with Betamethasone for lung maturation.
  HbA1C measurements from a blood draw of the patient.
Blood Glucose Level | One week after the medication with Betamethasone for lung maturation.
  Blood glucose level measurements from a blood draw of the patient.
Insulin level | One week after the medication with Betamethasone for lung maturation.
  Insulin level measurements from a blood draw of the patient.

OTHER OUTCOMES:
Age of the patient in years | At the day of the medication with betamethasone
  Age of the patient in years
Result of oral glucose tolerance test | The test will be carried out during pregnancy between 24+0 and 28+0 weeks of gestation
  Mandatory test in the Austrian Mother-Child-Pass. The data will be collected at the day of the medication with betamethasone.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Goebl, MD, Study Chair — AKH Vienna; Lara Linsenmeier, Student, Principal Investigator — Medical University of Vienna
Locations (1):
- AKH (General Hospital of) Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No